CLINICAL TRIAL: NCT04181424
Title: Lowering the Impact of Food Insecurity in African American Adults With Type 2 Diabetes Mellitus (LIFT-DM)
Acronym: LIFT-DM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Ehianu Egede, Professor & Chair, Department of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5R01MD013826 (NIH)
Record Dates: First submitted 2019-11-26; First posted 2019-11-29 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1- Diabetes Education Only (Active Comparator): Individuals assigned to this group will receive diabetes education and skills training but will not receive food supplementation.
  Interventions: Behavioral: Diabetes Education Only
- Group 2 - Diabetes Education Plus Monthly Food Vouchers (Experimental): Individuals assigned to this group will receive diabetes education and skills training and monthly food vouchers for use at local Farmer's markets mailed to their home.
  Interventions: Behavioral: Diabetes Education Plus Monthly Food Vouchers
- Group 3 - Diabetes Education Plus Monthly Stock Boxes (Experimental): Individuals assigned to this group will receive diabetes education and skills training and monthly stock boxes with diabetes appropriate food items mailed to their home.
  Interventions: Behavioral: Diabetes Education Plus Monthly Stock Boxes
- Group 4 -- Diabetes Education Plus Combination of Monthly Food (Experimental): Individuals assigned to this group will receive diabetes education and skills training, monthly food vouchers for use at local Farmer's markets mailed to their home, and monthly stock boxes with diabetes appropriate food items mailed to their home.
  Interventions: Behavioral: Diabetes Education Plus Combination of Monthly Food Vouchers and Stock Boxes

INTERVENTIONS:
Behavioral: Diabetes Education Plus Monthly Food Vouchers — Individuals assigned to this group will receive diabetes education and skills training and monthly food vouchers for use at local Farmer's markets mailed to their home.
  Arms: Group 2 - Diabetes Education Plus Monthly Food Vouchers
Behavioral: Diabetes Education Plus Combination of Monthly Food Vouchers and Stock Boxes — Individuals assigned to this group will receive diabetes education and skills training, monthly food vouchers for use at local Farmer's markets mailed to their home, and monthly stock boxes with diabetes appropriate food items mailed to their home.
  Arms: Group 4 -- Diabetes Education Plus Combination of Monthly Food
Behavioral: Diabetes Education Only — Individuals assigned to this group will receive diabetes education and skills training but will not receive food supplementation.
  Arms: Group 1- Diabetes Education Only
Behavioral: Diabetes Education Plus Monthly Stock Boxes — Individuals assigned to this group will receive diabetes education and skills training and monthly stock boxes with diabetes appropriate food items mailed to their home.
  Arms: Group 3 - Diabetes Education Plus Monthly Stock Boxes

SUMMARY:
The objective of this protocol is to answer the questions: 1) Within food supplementation options, are mailed stock boxes superior to food vouchers in terms of achieving glycemic control? 2) Is the combination of mailed stock boxes and food vouchers superior to either food supplementation option alone? 3) Does providing diabetes education in combination with food supplementation lead to improved clinical outcomes compared to education alone? To address this gap in the literature, we propose a randomized controlled trial to test the separate and combined efficacy of monthly food vouchers to farmers market and monthly mailed food stock boxes layered upon diabetes education in improving glycemic control in low income, food insecure, AAs with Type 2 Diabetes (T2DM) using a 2x2 factorial design.

DETAILED DESCRIPTION:
The overarching aim of this proposal is to conduct a 4-arm RCT to test the separate and combined efficacy of monthly food vouchers to farmers market and monthly mailed food stock boxes layered upon diabetes education in improving glycemic control in low income, food insecure, AAs with T2DM using a 2x2 factorial design. 300 patients will be randomly assigned to four groups of 75 patients each: 1) diabetes education alone; 2) diabetes education plus food vouchers; 3) diabetes education plus mailed stock boxes; and 4) diabetes education plus combined food vouchers and mailed stock boxes. Each patient will be followed for 12 months, with study assessments at baseline, 3, 6, and 12 months. Primary aim is efficacy of separate and combined interventions on HbA1c at 12 months post-randomization. Secondary aims are efficacy of separate and combined interventions on BP, LDL and QOL as well as cost-effectiveness at 12 months post-randomization.

Description of the LIFT-DM Intervention Group 1 - Diabetes Education Only: Individuals assigned to this group will receive diabetes education and skills training but will not receive food supplementation. Twelve 30-minute weekly sessions will be delivered via the telephone, with two 30-minute booster sessions at months 6 and 9.

Group 2 - Diabetes Education Plus Monthly Food Vouchers: Individuals assigned to this group will receive diabetes education and skills training and monthly food vouchers for use at local farmer's markets mailed to their home. Vouchers for $50 will be mailed monthly for 12 months.

Group 3 - Diabetes Education Plus Monthly Stock Boxes: Individuals assigned to this group will receive diabetes education and skills training and monthly stock boxes with diabetes appropriate food items mailed to their home. Stock boxes with foods valued at $50 will be mailed monthly for 12 months.

Group 4 - Diabetes Education Plus Combination of Monthly Food Vouchers and Stock Boxes: Individuals assigned to this group will receive diabetes education and skills training, monthly food vouchers for use at local farmer's markets mailed to their home, and monthly stock boxes with diabetes appropriate food items mailed to their home. Vouchers for $25 and stock boxes with food valued at $25 will be mailed monthly for 12 months. In essence, the combined group will still receive $50 worth of food supplementation monthly as combination of $25 vouchers and $25 mailed stock boxes.

ELIGIBILITY:
Inclusion Criteria: 1) age >=21 years; 2) self-report as African American/non-Hispanic Black; 3) screen positive for food insecurity over past 12-months using screening questionnaire; 4) clinical diagnosis of type 2 diabetes and HbA1c >=8% at the screening visit; 5) income <=133% of federal poverty level based on household income and size of household or Medicaid eligible; 6) able to communicate in English.

Exclusion Criteria: 1) Mental confusion on interview suggesting significant dementia; 2) Participation in other diabetes clinical trials; 3) Alcohol or drug abuse/dependency; 4) Active psychosis or acute mental disorder; and 5) Life expectancy <12 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Glycemic control (HbA1c) | 12-months post randomization
  Blood specimens (10cc of blood) will be obtained by trained phlebotomists or nurse for HbA1c.

SECONDARY OUTCOMES:
Quality of Life as measured by the SF-12 | 12-months post randomization
  The SF-12 (Ware 1996) is a valid and reliable instrument to measure functional status and reproduces 90% of the variance in PCS-36 and MCS-36 scores.
LDL-Cholesterol | 12-months post randomization
  About 10cc of blood will be drawn by trained phlebotomists and sent to the lab for LDL-Cholesterol.
Blood Pressure | 12-months post randomization
  Blood pressure readings will be obtained using automated BP monitors (OMRON IntelliSenseTM HEM-907XL). The device will be programmed to take 3 readings at 2-minute intervals, and give an average of the 3 BP readings.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard E Egede, MD, Principal Investigator — State University of New York at Buffalo; Rebekah J Walker, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- State University of New York at Buffalo, Buffalo, New York, United States

REFERENCES:
- [Background] Walker RJ, Knapp RG, Dismuke-Greer CE, Walker RE, Ozieh MN, Egede LE. Lowering the impact of food insecurity in African American adults with type 2 diabetes mellitus (LIFT-DM) - Study protocol for a randomized controlled trial. Contemp Clin Trials. 2020 Dec;99:106206. doi: 10.1016/j.cct.2020.106206. Epub 2020 Nov 7. PMID 33166622
- See also: Protocol paper — https://pubmed.ncbi.nlm.nih.gov/33166622/